CLINICAL TRIAL: NCT02100436
Title: A Phase II Open-Label Study in Healthy Pediatric Populations to Assess the Safety, Reactogenicity, and Immunogenicity of an Intramuscular Unadjuvanted Subvirion Monovalent Inactivated Influenza H3N2 Variant (H3N2v) Vaccine
Brief Title: Safety and Immunogenicity of a Monovalent Inactivated Influenza H3N2 Variant (H3N2v) Vaccine in Pediatric Populations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 12-0016; HHSN272200800002C
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2014-12-16

CONDITIONS: Influenza
Keywords: children; H3N2; H3N2v; influenza; pediatric; unadjuvanted; vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 3-8 years old (Experimental): up to 100 subjects receive 2 doses of H3N2v MIV, IM as 15mcg HA/0.5mL dose, 21 days apart.
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H3N2v A/Minnesota/11/2010 NYMC X-203
- Cohort 6-35 months old (Experimental): up to 100 subjects receive 2 doses of H3N2v MIV, intramuscularly (IM) as 7.5 micrograms (mcg) of hemagglutinin (HA)/0.25 milliliter (mL) dose, 21 days apart. up to 100 subjects receive 2 doses of H3N2v MIV, IM as 15mcg HA/0.5mL dose, 21 days apart.
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H3N2v A/Minnesota/11/2010 NYMC X-203
- Cohort 9-17 years old (Experimental): up tp 100 subjects receive 2 doses of H3N2v MIV, IM as 15mcg HA/0.5mL dose, 21 days apart.
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H3N2v A/Minnesota/11/2010 NYMC X-203

INTERVENTIONS:
Biological: Influenza Virus Vaccine, Monovalent A/H3N2v A/Minnesota/11/2010 NYMC X-203 — A unadjuvanted subvirion monovalent inactivated split influenza virus vaccine (H3N2v MIV) produced in eggs. Subjects are enrolled in 3 cohorts stratified by age. 6-35 month old subjects receive 2 doses of H3N2v MIV, intramuscularly (IM) as 7.5 micrograms (mcg) of hemagglutinin (HA)/0.25 milliliter (mL) dose, 21 days apart, or 2 doses of H3N2v MIV, IM as 15mcg HA/0.5mL dose, 21 days apart. 3-8 year old subjects and 9-17 year old subjects receive 2 doses of H3N2v MIV, IM as 15mcg HA/0.5mL dose, 21 days apart.

SUMMARY:
This is a Phase II open-label study in approximately 240, and up to 400, healthy males and non-pregnant females, aged 6 months to 17 years. This study is designed to assess the safety, reactogenicity, and immunogenicity of two doses administered intramuscularly approximately 21 days apart of an unadjuvanted subvirion monovalent inactivated influenza H3N2v vaccine manufactured by sanofi pasteur. Subjects will be stratified by age (approximately 60-100 subjects 6-35 months old, approximately 60-100 subjects 3-8 years old and approximately 60-100 subjects 9-17 years old) to receive 2 doses of vaccine, administered intramuscularly as 15mcg HA/0.5mL dose, approximately 21 days apart. In addition, approximately 60-100 subjects 6-35 months old will receive 2 doses of vaccine, administered intramuscularly as 7.5mcg HA/0.5mL dose, approximately 21 days apart. The duration of the study for each subject will be approximately 7 months.

DETAILED DESCRIPTION:
This is a Phase II open-label study in approximately 240 (up to 400) healthy males and non-pregnant females, 6 months to 17 years old, inclusive. This study is designed to assess the safety, reactogenicity, and immunogenicity of two doses administered intramuscularly approximately 21 days apart of an unadjuvanted subvirion monovalent inactivated influenza H3N2 variant (H3N2v) vaccine (MIV) manufactured by sanofi pasteur. Subjects will be stratified by age (approximately 120 (up to 200) subjects 6-35 months old, approximately 60 (up to 100) subjects 3-8 years old, and approximately 60 (up to 100) subjects 9-17 years old). Subjects in the 6-35 months old cohort will be randomized to receive either two doses of H3N2v MIV, administered intramuscularly as 7.5 micrograms (mcg) of hemagglutinin (HA)/0.25 milliliter (mL) dose (approximately 60 (up to 100) subjects), approximately 21 days apart, or two doses of H3N2v MIV, administered intramuscularly as 15mcg HA/0.5mL dose (approximately 60 (up to 100) subjects), approximately 21 days apart. All subjects in the 3-8 years old cohort and 9-17 years old cohort will receive two doses of H3N2v MIV, delivered intramuscularly as 15mcg HA/0.5mL dose, approximately 21 days apart. Subjects may receive licensed seasonal influenza vaccine prior to (>2 weeks if given the inactivated vaccine or >4 weeks if given the live, attenuated vaccine) the first H3N2v vaccination. Alternatively, subjects may receive licensed seasonal influenza vaccine at any time after completion of Visit 05 or following an early termination visit. Safety will be measured by the occurrence of solicited injection site and systemic reactogenicity from the time of each H3N2v vaccination through 7 days after each H3N2v vaccination. Unsolicited non-serious adverse events (AEs) will be collected from the time of the H3N2V vaccination (Day 0 (Visit 01)) through approximately 21 days after the last H3N2v vaccination (approximately Day 42 (Visit 05) for subjects who receive two H3N2v vaccinations; approximately Day 21 (Visit 03) for subjects who receive only one H3N2v vaccination). After approximately 21 days after the last H3N2v vaccination, non-serious AEs will be limited to new-onset chronic medical conditions, which will be documented through approximately 7 months after the first H3N2v vaccination (Visit 08). Serious adverse events (SAEs) will be collected from the time of the first H3N2v vaccination (Day 0 (Visit 01)) through approximately 7 months after the first H3N2v vaccination (Visit 08). Immunogenicity testing will include performing hemagglutination inhibition (HAI) and neutralizing (Neut) antibody assays on serum obtained prior to each H3N2v vaccination (Day 0 (Visit 01) and approximately Day 21 (Visit03)) and approximately 21 days after the second H3N2v vaccination (Visit 05).

ELIGIBILITY:
Inclusion Criteria:

1. Parent(s)/legal guardian(s) must provide written informed consent (parental permission) and subjects must provide written assent as appropriate for age per local IRB and 45 CFR 46 requirements prior to initiation of any study procedures. 2. Parent(s)/legal guardian(s) and subjects as appropriate must be willing and able to comply with planned study procedures and be available for all study visits. 3. Are males or non-pregnant females aged 6 months to 17 years old, inclusive. 4. Are in good health, as determined by medical history and targeted physical examination based on medical history. 5. Axillary temperature is less than 100°F, or oral temperature is less than 101°F. 6. Females of childbearing potential (status as determined by local IRB guidelines for minimum age requirements, and/or by occurrence of menarche and not having reached menopause >/=1 year or not having been surgically sterilized via tubal ligation, bilateral oophorectomy or hysterectomy) must agree to practice adequate contraception (abstinence from sexual intercourse with males, monogamous relationship with a vasectomized partner who was vasectomized at least 6 months prior to the subject receiving the first H3N2v vaccination, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices (IUDs), NuvaRing®, successful Essure® placement (permanent, non-surgical, non-hormonal sterilization) with documented confirmation test at least 3 months after the procedure, licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill"), and any other Food and Drug Administration (FDA) approved birth control method) for at least 30 days prior to the first H3N2v vaccination through at least 30 days after the last H3N2v vaccination. Method of contraception will be captured on the appropriate data collection form. 7. Females of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to each H3N2v vaccination.

Exclusion Criteria:

1. Have an acute illness, including an axillary temperature greater than or equal to 100°F or an oral temperature greater than or equal to 101°F, within 3 days prior to each H3N2v vaccination. 2. Have any condition that, in the opinion of the site principal investigator or appropriate sub-investigator, would place the subject at an unacceptable risk of injury, render them unable to meet the requirements of the protocol or confound the interpretation of results. 3. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months. 4. Have known active neoplastic disease or a history of any hematologic malignancy. 5. Have known HIV, hepatitis B, or hepatitis C infection. 6. Have a known allergy to eggs, egg or chicken protein, or other components of the H3N2v MIV (including octylphenol ethoxylate (Triton® X-100), gelatin, formaldehyde, and phosphate buffered saline). 7. Have a history of severe reactions following previous immunization with licensed influenza virus vaccines. 8. Have a history of Guillain-Barré Syndrome. 9. Have a history of alcohol or drug abuse in the past 5 years. 10. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other major psychiatric diagnosis or a static or progressive neurodevelopmental disorder (e.g. Cerebral palsy with mental retardation). 11. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years. 12. Have taken oral or parenteral corticosteroids of any dose within the past 4 weeks. 13. Have taken high-dose inhaled corticosteroids within the past 4 weeks. High dose defined as >840mcg/day (children 12-17 years of age) or >672mcg/day (children <12 years of age) of beclomethasone dipropionate CFC or equivalent. 14. Have used any topical steroid daily for more than 3 weeks within the past 3 months. 15. Received any licensed live vaccine within 4 weeks or any licensed inactivated vaccine within 2 weeks prior to the first H3N2v vaccination or planned receipt of any vaccine within 42 days after the first H3N2v vaccination. This is inclusive of licensed seasonal influenza vaccines and routine childhood immunizations provided outside the scope of this study.The initiation of this protocol does not take precedence over routine childhood immunizations. 16. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 3 months prior to each H3N2v vaccination. 17. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to the first H3N2v vaccination. 18. Are participating or plan to participate in another clinical trial with an interventional agent (licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication) during the 7-month study period. 19. Are enrolled or plan to enroll in another clinical trial that has a study intervention such as a drug, biologic, device, blood product, or medication that could interfere with the safety assessment of the investigational product at any time during the 7-month study period. 20. Participated in an influenza A/H3N2v vaccine study in the past in a group receiving vaccine (does not apply to documented placebo recipients) or have a history of A/H3N2v infection prior to enrollment. 21. Plan to travel outside the US (continental US, Hawaii and Alaska) in the time between the first H3N2v vaccination and 42 days after the first H3N2v vaccination. 22. Females who are breastfeeding or plan to breastfeed at any given time during the 7-month st udy period. 23. Occupational exposure to or substantial direct physical contact with pigs in the past year or during the 42 days after the first H3N2v vaccination. Casual contact with pigs at petting zoos or county or state fairs, for example,does not exclude subjects from study participation.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 270 (Actual)
Dates: Start 2014-06-11 (Actual); Primary Completion 2015-03-20 (Actual); Study Completion 2015-03-20 (Actual)

PRIMARY OUTCOMES:
Occurrence of H3N2v MIV-related serious adverse events from the time of the first H3N2v vaccination through approximately 7 months after the first H3N2v vaccination. | First vaccination (Day 0) through 7 months.
Occurrence of solicited injection site and systemic reactogenicity from the time of each H3N2v vaccination through 7 days after each H3N2v vaccination. | Through 7 days after each H3N2v vaccination.
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the H3N2v antigen contained in the H3N2v MIV following receipt of first dose of H3N2v MIV. | 6-35 months old and 3-8 year old cohorts, approximately 42 days. 9-17 years old cohort, approximately 21 days.
Percentage of subjects achieving seroconversion (defined as either pre-vacc. HAI titer < 1:10 and post-vacc. HAI titer >/=1:40 or pre-vacc. HAI titer >/=1:10 and minimum 4 fold rise in post-vacc. HAI antibody titer) following first dose of H3N2v MIV. | 6-35 months old and 3-8 years old cohorts, approximately 42 days. 9-17 years old cohort, approximately 21 days.

SECONDARY OUTCOMES:
Geometric Mean Titers of serum HAI and Neut antibody following receipt of each dose of H3N2v. | Baseline and approximately 21 days following receipt of each dose.
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the H3N2v antigen contained in the H3N2v MIV following receipt of the first dose of H3N2v MIV. | 6-35 months old and 3-8 years old cohorts, baseline and approximately 21 days. 9-17 years old cohort, baseline and approximately 42 days.
Percentage of subjects achieving a serum Neut antibody titer of 1:40 or greater against the H3N2v antigen contained in the H3N2v MIV following receipt of each dose of H3N2v MIV. | Baseline and approximately 21 days following receipt of each dose.
Percentage of subjects achieving seroconversion (defined as either pre-vacc. HAI titer < 1:10 and post-vacc. HAI titer >/=1:40 or pre-vacc. HAI titer >/=1:10 and a minimum 4 fold rise in post-vacc. HAI antibody titer)following first dose of H3N2v MIV. | 6-35 months old and 3-8 years old cohorts, approximately 21 days. 9-17 years old cohort, approximately 42 days.
Percentage of subjects achieving seroconversion (either pre-vacc. Neut titer < 1:10 and post-vacc. Neut titer >/=1:40 or pre-vacc. Neut titer >/=1:10 and minimum 4 fold rise in post-vacc. Neut antibody titer) following receipt of each dose of H3N2v MIV. | Approximately 21 days following receipt of each dose.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Children's Mercy Hospital and Clinics - Infectious Diseases, Kansas City, Missouri
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Duke Health Center at Roxboro, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas

REFERENCES:
- [Derived] Munoz FM, Anderson EJ, Bernstein DI, Harrison CJ, Pahud B, Anderson E, Creech CB, Berry AA, Kotloff KL, Walter EB, Atmar RL, Bellamy AR, Chang S, Keitel WA. Safety and immunogenicity of unadjuvanted subvirion monovalent inactivated influenza H3N2 variant (H3N2v) vaccine in children and adolescents. Vaccine. 2019 Aug 23;37(36):5161-5170. doi: 10.1016/j.vaccine.2019.07.085. Epub 2019 Jul 30. PMID 31375440